CLINICAL TRIAL: NCT05107115
Title: A Randomized, Double-blind, Placebo-controlled, Multi-center, Dose-ranging Phase 2 Study of Rilzabrutinib Followed by an Open-label Extension Phase in Patients With Moderate-to-severe Chronic Spontaneous Urticaria (CSU) Who Remain Symptomatic Despite the Use of H1 Antihistamine Treatment
Brief Title: Rilzabrutinib for the Treatment of Chronic Spontaneous Urticaria in Patients Who Remain Symptomatic Despite the Use of H1 Antihistamine
Acronym: RILECSU
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DRI17224; U1111-1263-4226 (Registry Identifier: ICTRP); DRI17224 (Other: Sanofi Identifier); 2021-002609-93 (EudraCT Number)
Record Dates: First submitted 2021-10-27; First posted 2021-11-04 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Chronic Spontaneous Urticaria
MeSH Terms: conditions — Chronic Urticaria

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Rilzabrutinib dose A (Experimental): dose A
  Interventions: Drug: rilzabrutinib
- Rilzabrutinib dose B (Experimental): dose B
  Interventions: Drug: rilzabrutinib
- Rilzabrutinib dose C (Experimental): dose C
  Interventions: Drug: rilzabrutinib
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: rilzabrutinib — Tablet, oral use
  Other Names: PRN1008/SAR444671
  Arms: Rilzabrutinib dose A; Rilzabrutinib dose B; Rilzabrutinib dose C
Drug: placebo — Tablet, oral use
  Arms: Placebo

SUMMARY:
The first phase of this study will be a parallel, 12-week treatment, Phase 2, double-blind, 4 arm study to assess the safety and effectiveness of 3 oral doses of SAR444671 (rilzabrutinib), i.e. dose A, B and C, compared with placebo for decreasing the frequency and severity of itch and urticaria in male and female participants aged 18 years inclusive or older with CSU.

After completion of the double-blind phase of the study, participants will be given the option of enrolling in the 40-week open label extension (OLE) phase of the study. Participants will receive open-label rilzabrutinib at dose C (the dose may be modified based on the 12-week safety and efficacy data). Due to the fact that some participants may be receiving rilzabrutinib for the first time, all participants will be monitored at Week 14, Week 16, Week 20, and Week 24. Afterwards, participants will be monitored at Week 36 and Week 52.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have a diagnosis of CSU refractory to H1-AH at the time of randomization
* Diagnosis of CSU ≥3 months prior to screening visit (Visit 1).
* The presence of itch and hives for ≥6 consecutive weeks at any time prior to screening visit (Visit 1) despite the use of H1-AH during this time period.
* Participants using a study defined H1-AH for CSU treatment. For participants on stable doses of non-study-approved H1-AH, investigators may switch participants to an equivalent dose of a study-approved H1-AH maintenance medication.
* Participants who are omalizumab naïve OR omalizumab-incomplete responders.
* Participants must be willing and able to complete a daily symptom e-diary for the duration of the study.
* During the 7 days before randomization: UAS7 ≥16 and ISS7 ≥8.
* Contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Exclusion Criteria:

* Clearly defined underlying etiology for CUs other than CSU (main manifestation being physical urticaria).
* Presence of skin morbidities other than CSU that may interfere with the assessment of the study outcomes.
* Participants with active atopic dermatitis (AD).
* Severe concomitant illness(es) that, in the Investigator's judgment, would adversely affect the patient's participation in the study.
* Known or suspected immunodeficiency, or otherwise recurrent infections of abnormal frequency or prolonged duration suggesting an immune compromised status, as judged by the Investigator.
* History of serious infections requiring intravenous (IV) therapy with the potential for recurrence (as judged by the Site Investigator) with less than 4 weeks interval between resolution of serious infection and first dose of study drug, or currently active moderate to severe infection at Screening (Grade 2 or higher), including active coronavirus disease 2019 (COVID-19).
* Live vaccine except Bacille Calmette Guerin-vaccination within 28 days prior to Day 1 or plan to receive one during the trial; Bacille Calmette Guerin-vaccination within 12 months prior to Screening.
* Active malignancy or history of malignancy within 5 years.
* Conditions that may predispose the participant to excessive bleeding
* Any participant with an uncontrolled disease state as judged by the Investigator, such as asthma, psoriasis, or inflammatory bowel disease, etc. that are typically treated with oral or parenteral corticosteroids
* Previous use of a BTK inhibitor.
* Has received any investigational drug (or is currently using an investigational device) within the 30 days before Day 1, or at least 5 times the respective elimination half-life time (whichever is longer).
* Previous exposure to another investigative drug for CSU.
* Positive for human immunodeficiency virus (HIV) antibody test.
* Presence of hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) with positive DNA test result at screening or within 3 months prior to the screening visit.
* Positive hepatitis C antibody test result at screening or within 3 months prior to the screening visit.
* Tuberculosis infection.
* Any of significant laboratory abnormalities and ECG findings at the screening visit.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2021-11-24 (Actual); Primary Completion 2023-07-19 (Actual); Study Completion 2024-04-23 (Actual)

PRIMARY OUTCOMES:
Change from baseline in weekly urticaria activity score (UAS7) at Week 12 (except US and US reference countries) | From baseline to Week 12
For US and US reference countries only: change from baseline in weekly itch severity score (ISS7) at Week 12 | From baseline to Week 12

SECONDARY OUTCOMES:
Change from baseline in UAS7 at Week 4 | From baseline to Week 4
Change from baseline in ISS7 at Week 12 (except US and US reference countries) | From baseline to Week 12
For US and US reference countries only: change from baseline in UAS7 at Week 12 | From baseline to Week 12
Change from baseline in weekly hives severity score (HSS7) at Week 12 | From baseline to Week 12
Proportion of participants with UAS7 ≤6 at Week 12 | At Week 12
Proportion of participants with UAS7 = 0 at Week 12 | At Week 12
Incidence of treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), adverse events of special interest (AESIs) and withdrawals due to TEAEs during the double-blind period and the open label extension | Until Week 52
Plasma PK concentrations of rilzabrutinib in participants with CSU | Until Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (128):
- Argentina (12):
  - Investigational Site Number : 0320006, CABA, Buenos Aires
  - Investigational Site Number :0320006, CABA, Buenos Aires
  - Investigational Site Number : 0320002, CABA, Buenos Aires
  - Investigational Site Number :0320002, CABA, Buenos Aires
  - Investigational Site Number : 0320004, Rosario, Santa Fe Province
  - Investigational Site Number : 0320005, Rosario, Santa Fe Province
  - Investigational Site Number :0320004, Rosario, Santa Fe Province
  - Investigational Site Number :0320005, Rosario, Santa Fe Province
  - Investigational Site Number : 0320003, Rosario, Santa Fe Province
  - Investigational Site Number :0320003, Rosario, Santa Fe Province
  - Investigational Site Number : 0320001, Buenos Aires
  - Investigational Site Number :0320001, Buenos Aires
- Canada (13):
  - Investigational Site Number :1240010, Calgary, Alberta
  - Investigational Site Number : 1240009, Red Deer, Alberta
  - Investigational Site Number :1240009, Red Deer, Alberta
  - Investigational Site Number : 1240005, Toronto, Ontario
  - Investigational Site Number :1240005, Toronto, Ontario
  - Investigational Site Number : 1240004, Toronto, Ontario
  - Investigational Site Number :1240004, Toronto, Ontario
  - Investigational Site Number : 1240006, Montreal, Quebec
  - Investigational Site Number :1240006, Montreal, Quebec
  - Investigational Site Number : 1240002, Trois-Rivières, Quebec
  - Investigational Site Number :1240002, Trois-Rivières, Quebec
  - Investigational Site Number : 1240003, Québec
  - Investigational Site Number :1240003, Québec
- Chile (7):
  - Investigational Site Number : 1520004, Osorno, Los Lagos Region
  - Investigational Site Number :1520004, Osorno, Los Lagos Region
  - Investigational Site Number : 1520001, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number :1520001, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number :1520003, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520002, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number :1520002, Santiago, Reg Metropolitana de Santiago
- Germany (8):
  - Investigational Site Number :2760002, Berlin
  - Investigational Site Number : 2760002, Berlin
  - Investigational Site Number : 2760001, Dresden
  - Investigational Site Number :2760001, Dresden
  - Investigational Site Number : 2760005, Kiel
  - Investigational Site Number :2760005, Kiel
  - Investigational Site Number : 2760004, Mainz
  - Investigational Site Number :2760004, Mainz
- Greece (8):
  - Investigational Site Number : 3000001, Athens
  - Investigational Site Number :3000001, Athens
  - Investigational Site Number : 3000002, Athens
  - Investigational Site Number :3000002, Athens
  - Investigational Site Number : 3000004, N. Efkarpia
  - Investigational Site Number :3000004, N. Efkarpia
  - Investigational Site Number : 3000003, Thessaloniki
  - Investigational Site Number :3000003, Thessaloniki
- Italy (7):
  - Investigational Site Number : 3800001, Milan, Lombardy
  - Investigational Site Number :3800001, Milan, Lombardy
  - Investigational Site Number :3800004, Milan, Lombardy
  - Investigational Site Number : 3800002, Ancona
  - Investigational Site Number :3800002, Ancona
  - Investigational Site Number : 3800005, Catania
  - Investigational Site Number :3800005, Catania
- Japan (14):
  - Investigational Site Number :3920004, Nagoya, Aichi-ken
  - Investigational Site Number : 3920005, Chikushino-shi, Fukuoka
  - Investigational Site Number :3920005, Chikushino-shi, Fukuoka
  - Investigational Site Number : 3920002, Sapporo, Hokkaido
  - Investigational Site Number :3920002, Sapporo, Hokkaido
  - Investigational Site Number : 3920001, Sagamihara-shi, Kanagawa
  - Investigational Site Number :3920001, Sagamihara-shi, Kanagawa
  - Investigational Site Number : 3920007, Yokohama, Kanagawa
  - Investigational Site Number :3920007, Yokohama, Kanagawa
  - Investigational Site Number : 3920006, Izumo-shi, Shimane
  - Investigational Site Number :3920006, Izumo-shi, Shimane
  - Investigational Site Number : 3920003, Tachikawa-shi, Tokyo
  - Investigational Site Number :3920003, Tachikawa-shi, Tokyo
  - Investigational Site Number : 3920004, Nagoya
- Netherlands (4):
  - Investigational Site Number : 5280002, Rotterdam
  - Investigational Site Number :5280002, Rotterdam
  - Investigational Site Number : 5280001, Utrecht
  - Investigational Site Number :5280001, Utrecht
- Poland (15):
  - Investigational Site Number :6160007, Wroclaw, Lower Silesian Voivodeship
  - Investigational Site Number : 6160007, Wroclaw, Lower Silesian Voivodeship
  - Investigational Site Number : 6160001, Gdansk, Pomeranian Voivodeship
  - Investigational Site Number :6160001, Gdansk, Pomeranian Voivodeship
  - Investigational Site Number : 6160009, Gdansk, Pomeranian Voivodeship
  - Investigational Site Number :6160009, Gdansk, Pomeranian Voivodeship
  - Investigational Site Number : 6160008, Krakow
  - Investigational Site Number :6160008, Krakow
  - Investigational Site Number : 6160004, Krakow
  - Investigational Site Number :6160004, Krakow
  - Investigational Site Number :6160003, Krakow
  - Investigational Site Number : 6160005, Lodz
  - Investigational Site Number :6160005, Lodz
  - Investigational Site Number : 6160006, Wroclaw
  - Investigational Site Number :6160006, Wroclaw
- Russia (9):
  - Investigational Site Number : 6430005, Moscow
  - Investigational Site Number :6430005, Moscow
  - Investigational Site Number :6430006, Moscow
  - Investigational Site Number : 6430002, Moscow
  - Investigational Site Number :6430002, Moscow
  - Investigational Site Number :6430003, Saint Petersburg
  - Investigational Site Number :6430004, Smolensk
  - Investigational Site Number : 6430001, Stavropol
  - Investigational Site Number :6430001, Stavropol
- South Korea (9):
  - Investigational Site Number : 4100002, Busan, Busan
  - Investigational Site Number :4100002, Busan, Busan
  - Investigational Site Number : 4100005, Ansan-si, Gyeonggi-do
  - Investigational Site Number :4100005, Ansan-si, Gyeonggi-do
  - Investigational Site Number :4100001, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100003, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number :4100003, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100004, Yeongdeunpo-gu, Seoul-teukbyeolsi
  - Investigational Site Number :4100004, Yeongdeunpo-gu, Seoul-teukbyeolsi
- Spain (14):
  - Investigational Site Number : 7240004, Seville, Andalusia
  - Investigational Site Number :7240004, Seville, Andalusia
  - Investigational Site Number : 7240001, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number :7240001, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240008, Barcelona / Sabadell, Catalunya [Cataluña]
  - Investigational Site Number :7240008, Barcelona / Sabadell, Catalunya [Cataluña]
  - Investigational Site Number :7240007, Pozuelo de Alarcón, Madrid
  - Investigational Site Number : 7240006, Pamplona, Navarre
  - Investigational Site Number :7240003, Pamplona, Navarre
  - Investigational Site Number :7240006, Pamplona, Navarre
  - Investigational Site Number : 7240005, Alicante
  - Investigational Site Number :7240005, Alicante
  - Investigational Site Number : 7240002, Córdoba
  - Investigational Site Number :7240002, Córdoba
- Taiwan (8):
  - Investigational Site Number : 1580002, Hsinchu
  - Investigational Site Number :1580002, Hsinchu
  - Investigational Site Number : 1580004, Kaohsiung City
  - Investigational Site Number :1580004, Kaohsiung City
  - Investigational Site Number : 1580003, Taichung
  - Investigational Site Number :1580003, Taichung
  - Investigational Site Number : 1580001, Taipei
  - Investigational Site Number :1580001, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Gimenez-Arnau A, Ferrucci S, Ben-Shoshan M, Mikol V, Lucats L, Sun I, Mannent L, Gereige J. Rilzabrutinib in Antihistamine-Refractory Chronic Spontaneous Urticaria: The RILECSU Phase 2 Randomized Clinical Trial. JAMA Dermatol. 2025 Jul 1;161(7):679-687. doi: 10.1001/jamadermatol.2025.0733. PMID 40266575